CLINICAL TRIAL: NCT02156193
Title: Effect of Prophylactic Clip Application for the Prevention of Postpolypectomy Bleeding in Large Pedunculated Colonic Polyps: a Randomized, Controlled Trial
Brief Title: Effect of Prophylactic Clip Application for the Prevention of Postpolypectomy Bleeding in Pedunculated Colonic Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jeong-Seon Ji, Dr, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clip control
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic clip (Experimental): Before conventional snare polypectomy, hemoclips will be applied on the base of stalk.
  Interventions: Procedure: Prophylactic clip
- No prophylactic management (Active Comparator): Conventional snare polypectomy will be performed without any preventive management.
  Interventions: Procedure: No prophylactic management

INTERVENTIONS:
Procedure: Prophylactic clip — Prophylactic clipping
  Arms: Prophylactic clip
Procedure: No prophylactic management — No prophylaxis
  Arms: No prophylactic management

SUMMARY:
Although endoscopic colonic polypectomy has been an established procedure for two decades, the risk of bleeding is still higher after resecting of pedunculated polyps, because of the presence of a large artery in the stalk. Preventive methods such as endoloop and epinephrine injection have been proposed in the management of postpolypectomy bleeding in large colonic polyps. For prophylactic clip, there was no randomized controlled study assessing the efficacy in the prevention of postpolypectomy bleeding for the large pedunculated polyps. So the investigators designed a randomized controlled trial to confirm the efficacy of application of prophylactic clip in the prevention of postpolypectomy bleeding in large polyps.

DETAILED DESCRIPTION:
Patients who had pedunculated colorectal polyps with heads larger than 10 mm and stalks larger than 5 mm in diameter were included. In clip group, hemoclips were applied to the base of the stalk, followed by conventional snare polypectomy. In conventional group, conventional snare polypectomy was done without any preventive management. Immediate and delayed bleeding complications were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pedunculated colorectal polyps, the heads of which were larger than 10mm and the stalk of which were large than 5 mm in diameter, were included.

Exclusion Criteria:

* bleeding tendency, poor preparation, sessile polyp

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Postpolypectomy bleeding | 1 month
  Immediate and delayed postpolypectomy bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Seon Ji, Dr, Principal Investigator — Incheon St. Mary's Hospital, The Catholic University of Korea
Locations (1):
- Incheon St. Mary's Hospital, The Catholic University of Korea, Incheon, South Korea

REFERENCES:
- [Derived] Gweon TG, Lee KM, Lee SW, Kim DB, Ji JS, Lee JM, Chung WC, Paik CN, Choi H. Effect of prophylactic clip application for the prevention of postpolypectomy bleeding of large pedunculated colonic polyps: a randomized controlled trial. Gastrointest Endosc. 2021 Jul;94(1):148-154. doi: 10.1016/j.gie.2020.12.040. Epub 2021 Jan 5. PMID 33417897